CLINICAL TRIAL: NCT04953715
Title: Microbiome and Immunosuppression: The Mission Study
Acronym: MISSION
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-0273; R01AI140303 (NIH); "MISSION" study (Other: Hennepin Healthcare Research Institute)
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant
Keywords: transplant; kidney; Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from whole blood, microbiome stool and oral samples will be processed and stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 - This is a multicenter microbiome and pharmacokinetic study.: A prospective, observational microbiome study of adult kidney transplant recipients receiving mycophenolate mofetil and tacrolimus maintenance immunosuppression. Participants will be studied post-transplant for mycophenolate pharmacokinetics and microbiome samples collected. Clinically measured tacrolimus trough concentrations will also be evaluated. Associations among mycophenolic acid enterohepatic recycling and metabolite formation, tacrolimus troughs, immunosuppression adverse effects, diarrhea and microbiome will be studied. To assess the relationship between kidney graft outcomes and stool, oral, nasal and urine microbiome diversity. To assess the relationship between transplant graft outcomes and urinary transcriptome.
  Interventions: Other: collection of body microbiome

INTERVENTIONS:
Other: collection of body microbiome — A prospective, observational microbiome study of adult kidney transplant recipients receiving mycophenolate mofetil and tacrolimus maintenance immunosuppression. Participants will be studied post-transplant for mycophenolate pharmacokinetics and microbiome samples collected. Clinically measured tacrolimus trough concentrations will also be evaluated. Associations among mycophenolic acid enterohepatic recycling and metabolite formation, tacrolimus troughs, immunosuppression adverse effects, diarrhea and microbiome will be studied.

SUMMARY:
The purpose of this research is to study immunosuppression drugs, certain foods, and how they can change the microbiome (the natural microorganisms inside the body) of the individual taking the immunosuppressive medications. The study team wants to study how the microbiome affects how the body processes the transplant medication.

DETAILED DESCRIPTION:
Immunosuppression drugs, like antibiotics and certain foods, can change the microbiome (the natural micro-organisms inside the body) of the individual taking the drug. The study team wants to study what impact these changes to the microbiome have on the individual. The study team is specifically interested in how these changes to the microbiome may change the metabolism (breakdown) and action of medications. It is already known that individual genetics impact the metabolism, absorption, and toxicities of some medications. It is suspected that the microbiome will have similar impacts on medications. With a better understanding of how individual microbiome impacts immunosuppressant medications used to help transplant recipients from rejecting their new organs, providers can more accurately prescribe and dose these medications to better treat and care for transplant patients and their organs.

It is expected that participants will be in this research study for up to 12 years. There will be periods of time that requires active participation (visits) and periods of time that will be more passive participation (allowing study staff to follow-up with medical records for outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing kidney transplant
* Male or female at least 18 years of age at time of enrollment
* Will or have received a living or deceased donor kidney transplant
* Planned post-transplant immunosuppression regimen of mycophenolate mofetil dosed every 12 hours (Cellcept or generic) and immediate release tacrolimus dosed twice daily with trough concentration monitoring (generic or brand formulation).
* Able and willing to complete study-related procedures and visits
* Signs written informed consent

Exclusion Criteria:

* Recipient of a previous non-kidney transplant
* Subject is a multi-organ transplant recipient
* Presence of active gastroparesis, and documented in the medical record
* Liver dysfunction (total bilirubin >2x upper limit of normal) within 2 months of enrollment
* Patients who take medications that significantly inhibit uridine 5'-diphosphate glucuronosyltransferase (UGT) enzymes.
* Patients who take medications that significantly inhibit or induce the biliary transporters
* Patient is known to be HIV positive
* Pregnant or nursing (lactating) women
* Non-English speaking
* Patients who have undergone bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults kidney transplant recipients with a planned immunosuppression regimen of mycophenolate mofetil dosed every 12 hours and immediate release tacrolimus dosed twice daily.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
To assess the relationship between transplant graft outcomes and urinary transcriptome. | 5 years
  The gut microbiome has been implicated in the Stool from tx recipients with diarrhea is often sent for testing of potential pathogenic organisms. polymerase chain reaction (PCR)- based approaches to identify etiology of post-tx diarrhea only tests for a limited number of organisms.
To assess the relationship between kidney graft outcomes and stool, oral, nasal, and urine microbiome diversity. | 5 years
  The gut microbiome has been implicated in the variability in metabolism of drugs with specific microbial species being associated with direct and indirect effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Israni, MD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - HCMC, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed ME, Saqr A, Onyeaghala G, Remmel RP, Staley C, Dorr CR, Teigen L, Guan W, Vo D, El-Rifai R, Oetting WS, Matas AJ, Israni AK, Jacobson PA. A Mycophenolate Pharmacokinetic Study with New Insights into Enterohepatic Recirculation in Kidney Transplant Recipients. Clin Pharmacokinet. 2026 Feb 6. doi: 10.1007/s40262-025-01611-3. Online ahead of print. PMID 41649771
- [Derived] Mohamed ME, Saqr A, Onyeaghala G, Remmel RP, Staley C, Dorr CR, Teigen L, Guan W, Madden H, Munoz J, Sanchez B, Vo D, El-Rifai R, Oetting WS, Matas AJ, Israni AK, Jacobson PA. Simultaneous Prediction of Area Under the Curves of Mycophenolic Acid and Its Metabolites and Enterohepatic Recirculation in Kidney Transplant Recipients. Ther Drug Monit. 2025 Dec 1;47(6):799-808. doi: 10.1097/FTD.0000000000001336. Epub 2025 Apr 30. PMID 40315256
- [Derived] Mohamed ME, Saqr A, Al-Kofahi M, Onyeaghala G, Remmel RP, Staley C, Dorr CR, Teigen L, Guan W, Madden H, Munoz J, Vo D, Sanchez B, El-Rifai R, Oetting WS, Matas AJ, Israni AK, Jacobson PA. Limited Sampling Strategies Fail to Accurately Predict Mycophenolic Acid Area Under the Curve in Kidney Transplant Recipients and the Impact of Enterohepatic Recirculation. Ther Drug Monit. 2025 Feb 1;47(1):174-182. doi: 10.1097/FTD.0000000000001248. Epub 2024 Jul 23. PMID 39047238